CLINICAL TRIAL: NCT04002466
Title: Evaluation of Dietary Iron Intake, Anemia, and Iron Status Among Men, Women, and Children in Ethiopia
Brief Title: Anemia Etiology Evaluation in Ethiopia
Acronym: AnemEE
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Addis Continental Institute of Public Health (Other)
Responsible Party: Principal Investigator, Wafaie Fawzi, Professor of Nutrition, Epidemiology, and Global Health, Harvard School of Public Health (HSPH)
Other Study IDs: OPP1179606
Record Dates: First submitted 2019-06-21; First posted 2019-06-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Risk Factors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children (6-59 months)
  Interventions: Other: Risk factors for anemia
- Women of Reproductive Age (15-49 years)
  Interventions: Other: Risk factors for anemia
- Adult Men (15-49 years)
  Interventions: Other: Risk factors for anemia

INTERVENTIONS:
Other: Risk factors for anemia — Diet, iron, vitamin B12, folate, inflammation, soil transmitted helminth infection, malaria, other morbidities and other health/nutrition/sociodemographic factors

SUMMARY:
The AnemEE study is a population-based anemia etiology survey in six regions of Ethiopia. The primary aim of the study is to evaluate the relative contribution of risk factors for anemia among children, women of reproductive age, and adult men. The study data are intended to inform evidence-based decision-making on anemia control interventions.

DETAILED DESCRIPTION:
The AnemEE study is a population-based cross-sectional survey of children (6-59 months), adult women of reproductive age (15-49 years) and adult males (15-49 years) in six regions of Ethiopia (Afar, Amhara, Tigray, Oromia, Southern Nations, Nationalities and Peoples' Region and Addis Ababa). The study will enroll approximately 5,100 participants and will be conducted in two survey rounds; one survey round in the Belg season and one survey round in the Meher season. All participants will have hemoglobin assessed and will have standardized questionnaires administered to assess sociodemographic, diet, morbidity, and other health/nutrition factors. All participants will also have assessments of anthropometric measures, malaria, and soil transmitted helminth infection. A subset of participants will also have serum ferritin, CRP, AGP, vitamin B12, and folate concentrations assessed. The study data will be used to determine the relative contributions of risk factors for anemia.

ELIGIBILITY:
Inclusion Criteria:

1. Women of reproductive age

   * Female living in a selected household that has a woman 15-49 years of age
   * Aged 15-49 years
2. Adult Men

   * Male living in a selected household that has a woman 15-49 years of age
   * Aged 15-49 years
3. Children

   * Male or female child living in a selected household that has a woman 15-49 years of age
   * Aged 6-59 months

Exclusion Criteria:

* Does not provide informed consent

Ages: 6 Months to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children (6-59 months); Women of reproductive age (15-49 years); Adult men (15-49 years)
Sampling Method: Probability Sample
Enrollment: 5114 (Actual)
Dates: Start 2019-01-27 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Anemia | One day
  Hemoglobin concentration by sex and age (<11 g/dL for children; Hb <12 g/dL for non-pregnant adult women, <13 g/dL for adult men). Hemoglobin concentrations will be adjusted for altitude and smoking status.

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MBBS, DrPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Addis Continental Institute of Public Health, Addis Ababa, Ethiopia

REFERENCES:
- [Derived] Tadesse AW, Hemler EC, Andersen C, Passarelli S, Worku A, Sudfeld CR, Berhane Y, Fawzi WW. Anemia prevalence and etiology among women, men, and children in Ethiopia: a study protocol for a national population-based survey. BMC Public Health. 2019 Oct 24;19(1):1369. doi: 10.1186/s12889-019-7647-7. PMID 31651278